CLINICAL TRIAL: NCT02497313
Title: Effect of Metformin and Cholecystokinin-mediated Gallbladder Emptying on GLP-1 Secretion in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Andreas Brønden, MD, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: H-15007280
Record Dates: First submitted 2015-07-09; First posted 2015-07-14 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sodium Chloride; Cholecystokinin; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo+Placebo (Placebo Comparator): Oral ingestion of metformin placebo combined with intravenous infusion of isotonic saline.
  Interventions: Drug: Isotonic saline; Drug: Metformin placebo
- Placebo+Cholecystokinin (Active Comparator): Oral ingestion of metformin placebo combined with intravenous infusion of cholecystokinin.
  Interventions: Drug: Metformin placebo; Drug: Cholecystokinin
- Metformin+Placebo (Active Comparator): Oral ingestion of metformin combined with intravenous infusion of isotonic saline.
  Interventions: Drug: Isotonic saline; Drug: Metformin
- Metformin+Cholecystokinin (Active Comparator): Oral ingestion of metformin combined with intravenous infusion of cholecystokinin.
  Interventions: Drug: Cholecystokinin; Drug: Metformin

INTERVENTIONS:
Drug: Isotonic saline
  Arms: Metformin+Placebo; Placebo+Placebo
Drug: Metformin placebo
  Arms: Placebo+Cholecystokinin; Placebo+Placebo
Drug: Cholecystokinin
  Arms: Metformin+Cholecystokinin; Placebo+Cholecystokinin
Drug: Metformin
  Arms: Metformin+Cholecystokinin; Metformin+Placebo

SUMMARY:
Accumulating evidence suggests that bile acids in our intestines may constitute essential components in the complex mechanisms regulating gut hormone secretion and glucose homeostasis. Thus, it is likely that modification of the enterohepatic circulation of bile acids can lead to changes in gut hormone secretion and consequently affect glucose homeostasis.

The current study is a human interventional randomized controlled cross-over study including four study days for each participant. Metformin will be applied as a tool to reduce bile acid reuptake in the small intestine; thereby increasing bile acid concentration in the more distal parts of the gut where GLP-1-secreting L cell are abundant. Interestingly, metformin has been shown to reduce the active reabsorption of bile acids in the ileum and cause increased faecal elimination of bile acids. Clinical data has suggested that metformin causes an increase in the postprandial secretion of GLP-1 in humans including patients with type 2 diabetes. Intravenous infusion of cholecystokinin will be used to elicit gallbladder contraction and emptying. The aim is to examine how (and if) modification of bile acid reabsorption can influence postprandial glucagon-like peptide-1 (GLP-1) secretion and glucose homeostasis in patients with type 2 diabetes.

The investigators hypothesize that higher luminal concentrations of bile acids in the distal gut will elicit changes in gut hormone secretion. The current study will help to clarify this hypothesis and improve our general understanding of the association between bile acid circulation and signalling, gut hormone secretion and glucose metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes for at least 3 months (diagnosed according to the criteria of the World Health Organization (WHO))
* Men and postmenopausal women
* Metformin applied as the only anti-diabetic drug
* Caucasian ethnicity
* Normal haemoglobin
* BMI >23 kg/m2 and <35 kg/m2
* Informed and written consent

Exclusion Criteria:

* Liver disease (alanine aminotransferase (ALAT) and/or serum aspartate aminotransferase (ASAT) >2 times normal values) or history of hepatobiliary disorder
* Gastrointestinal disease, previous intestinal resection, cholecystectomy or any major intra-abdominal surgery
* Nephropathy (serum creatinine >150 µM and/or albuminuria)
* Hypo- and hyperthyroidism
* Hypo- and hypercalcaemia
* Hypo- and hyperphosphataemia
* Active or recent malignant disease
* Treatment with medicine that cannot be paused for 12 hours
* Treatment with oral anticoagulants
* Any treatment or condition requiring acute or sub-acute medical or surgical intervention
* Any condition considered incompatible with participation by the investigators

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-07; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Glucagon-like peptide-1 (GLP-1): Incremental and total area under the Concentration-Time Curve | -30, -15, 0, 10, 20, 30, 45, 60, 90, 120, 180, 240 min on study days 1-4
  Incremental and total area under the Concentration-Time Curve (AUC 0-240 min)

SECONDARY OUTCOMES:
Responses of various other gut hormones: Incremental and total area under the Concentration-Time Curve | -30, -15, 0, 10, 20, 30, 45, 60, 90, 120, 180, 240 min on study days 1-4
  Incremental and total area under the Concentration-Time Curve (AUC 0-240 min)
Blood analysis of paracetamol as an assessment of gastric emptying | -30, -15, 0, 10, 20, 30, 45, 60, 90, 120, 180, 240 min on study days 1-4
  Assessment of gastric emptying
Indirect calorimetry: Basal metabolic rate | -30 min to 240 min
  Basal metabolic rate
Gallbladder volume as assessed by Ultrasound measurements | -30 min to 240 min
  Gallbladder volume
Appetite as assessed by Visual analog scale score | -30 min to 240 min
  Appetite

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Brønden, MD, Principal Investigator — PhD student
Locations (1):
- Center for Diabetes Research, Herlev-Gentofte Hospital, Hellerup, Denmark

REFERENCES:
- [Derived] Bronden A, Alber A, Rohde U, Rehfeld JF, Holst JJ, Vilsboll T, Knop FK. Single-Dose Metformin Enhances Bile Acid-Induced Glucagon-Like Peptide-1 Secretion in Patients With Type 2 Diabetes. J Clin Endocrinol Metab. 2017 Nov 1;102(11):4153-4162. doi: 10.1210/jc.2017-01091. PMID 28938439